CLINICAL TRIAL: NCT00726960
Title: Modulation of Opiate Reward by NK1 Antagonism: A Laboratory-Based Proof of Concept Study
Brief Title: Ability of Aprepitant to Block Opioid Reward in Non-Dependent Opiate Abusers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Ministry of Health and Social Affairs, Sweden (Other Government); County of Stockholm (Unknown)
Responsible Party: Markus Heilig, MD, PhD, Karolinska Universitetssjukhuset
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Aprepitant 1
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Opioid-Related Disorders; Heroin Dependence; Substance-Related Disorders
Keywords: Heroin abuse; Opioids; Opiates; Substance abuse; Addiction
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence; Substance-Related Disorders; Behavior, Addictive | interventions — Aprepitant; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aprepitant
  Interventions: Drug: aprepitant
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Pseudo-placebo - buprenorphine

INTERVENTIONS:
Drug: aprepitant — Oral, 125 mg once daily for one week
  Other Names: Emend
  Arms: 1
Drug: Pseudo-placebo - buprenorphine — Randomized to receive either 8 mg sublingual tablets or 0.4 mg sublingual tablets
  Other Names: Subutex
  Arms: 2

SUMMARY:
The objective of this study is to determine whether aprepitant blocks the opiate reward system in non-dependent opiate abusers, indicating its potential as a safe, non-addictive first line therapy for early heroin abuse.

DETAILED DESCRIPTION:
This initial proof-of-concept study focuses on evaluating whether an NK1 antagonist, aprepitant, can block opiate reward in non-dependent opiate experienced volunteers in response to a standard opiate challenge. Sixty subjects will be included in a randomized controlled study. Following a training challenge session, they will receive 1 week treatment with aprepitant or matching placebo, followed by a challenge session during which subjective and physiological responses to the opiate partial agonist buprenorphine will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 50
* Current opiate use, without dependence

Exclusion Criteria:

* Clinical diagnosis of opiate dependence
* Positive urine screen for opiates on day of challenge sessions
* Meet diagnostic criteria for any other substance abuse disorder except nicotine within the last 12 months.
* Any ongoing prescription medication other than oral contraceptives or hormone replacement
* Any serious medical condition which in the judgment of the investigators makes administration of opiates medically inappropriate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be self-reported pleasurable opiate effect. | One week

SECONDARY OUTCOMES:
The secondary outcome will be physiological opiate responses. | One week

CONTACTS AND LOCATIONS:
Overall Officials: Markus Heilig, MD, PhD, Principal Investigator — Karolinska University Hospital; Johan Kakko, MD, Study Director — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm, Sweden